CLINICAL TRIAL: NCT05709457
Title: Long Term Effects of an Intervention on Maternal Behavior, Child Health, and Community Influence
Brief Title: Long Term Effects Of a Maternal Cash Transfer Experiment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HD102412 (NIH)
Record Dates: First submitted 2022-10-19; First posted 2023-02-02 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maternal Health Services; Outcome Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCT Participants (Experimental): Women and children who participated in the earlier study.
  Interventions: Behavioral: Cash transfer in prior study
- Non-RCT participants (No Intervention): Women and children in the same communities included in the earlier study who did not participate in that study.

INTERVENTIONS:
Behavioral: Cash transfer in prior study — Women were offered a cash transfer conditional on attending prenatal and postnatal visits and delivering in a facility
  Arms: RCT Participants

SUMMARY:
This is a follow-on study to a cluster randomized trial of maternal conditional incentives conducted in Nigeria. This study found that cash transfers, conditional on women obtaining facility-based prenatal, delivery, and postnatal care, resulted in large, significant effects on maternal and child outcomes (NICHD R01HD083444). This study will answer additional key policy questions. First, are the effects on maternal behavior temporary, or do they result in more sustained behavior change? Second, do measured short run (SR) child health effects persist over the long run? Third, did the program generate spillovers?

DETAILED DESCRIPTION:
This study will build on what the study investigators learned from the RCT and extend it in novel directions. Research assistants will return to the study communities approximately 5 years after enrollment in the RCT to collect data on utilization of maternal health care services for births to the trial participants after the intervention, and on long run child health outcomes including child weight and height. The research assistants will also collect data on the birth outcomes of non-incentivized childbearing women in the study clusters. Data will be collected through in-person surveys of study participants.

This study will provide valuable new evidence about the indirect and long run effects of demand-side incentives. This is of critical importance because accounting for only the direct effects may severely underestimate the full effect of the program.

ELIGIBILITY:
Inclusion Criteria for Households:

* Resident in a community included in the RTC

Exclusion Criteria for Households:

* None

Inclusion Criteria for Women:

* Women must have participated in an earlier randomized trial of conditional incentives OR
* They did not take part in the earlier trial but are resident in clusters that participated in the earlier trial and have given birth since 2018

Exclusion Criteria for Women:

-

Ages: 13 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 21000 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of births that take place in a health facility | 4-5 years after RCT enrollment
  Proportion of births that take place in a health facility
Proportion of women that attended prenatal care during pregnancy | 4-5 years after RCT enrollment
  Proportion of women that attended prenatal care during pregnancy
Child survival | 4-5 years after RCT enrollment
  Probability that child is alive
Child health utilization | 4-5 years after RCT enrollment
  Proportion of children taken to a health facility for care when sick
Proportion of children receiving recommended immunizations | 4-5 years after RCT enrollment
  Proportion of children receiving recommended immunizations

SECONDARY OUTCOMES:
Maternal health | 4-5 years after RCT enrollment
  Self-rated health
Child weight | 4-5 years after RCT enrollment
  Child weight measured at visit
Child height | 4-5 years after RCT enrollment
  Child height measured at visit
Birth outcome | 4-5 years after RCT enrollment
  Probability of a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Okeke, MD, PhD, Principal Investigator — RAND
Locations (1):
- Amino Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared after results are published.
Supporting Information: Analytic Code